CLINICAL TRIAL: NCT03780244
Title: A Randomized, Evaluator-blinded, Multi-center Study to Evaluate the Safety and Effectiveness of Sculptra Aesthetic for Correction of Nasolabial Folds.
Brief Title: Safety and Effectiveness of Sculptra Aesthetic for Correction of Nasolabial Folds.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43USSA1705
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Results first posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: Nasolabial Folds

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Investigational Study Product (Experimental): Injection with Sculptra Aesthetic reconstituted with 8ml Sterile Water for Injection (SWFI)
  Interventions: Device: Sculptra Aesthetic 8ml
- Reference Product (Active Comparator): Injection with Sculptra Aesthetic reconstituted with 5ml SWFI
  Interventions: Device: Sculptra Aesthetic 5ml

INTERVENTIONS:
Device: Sculptra Aesthetic 8ml — Treatment of nasolabial folds
  Arms: Investigational Study Product
Device: Sculptra Aesthetic 5ml — Treatment of nasolabial folds
  Arms: Reference Product

SUMMARY:
This study has been designed to evaluate the safety of Sculptra Aesthetic as a single regimen for correction of Nasolabial Fold (NLF) contour deficiencies after changes in reconstitution and injection procedures compared to the approved label.

ELIGIBILITY:
Inclusion Criteria:

* Intent to undergo correction of both left and right NLFs with a Wrinkle Assessment Scale (WAS) score of greater than or equal to 2 (shallow wrinkles) to less than or equal to 4 (deep wrinkles) as assessed on Day 1 (and also at screening, if screening was performed prior to Day 1) by the Blinded Evaluator. A one grade difference between sides is allowed at inclusion.

Exclusion Criteria:

* Previous tissue augmenting therapy, contouring or revitalization treatment in or near the treatment area with any filler prior to Baseline visit.

  1. Collagen, Hyaluronic Acid- 12 months
  2. Calcium Hydroxyapatite (CaHa), Poly-L-lactic Acid (PLLA) or permanent (non-biodegradable)- Prohibited
* Known/previous allergy or hypersensitivity to any of the Sculptra Aesthetic constituents.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Galderma Study Site, Scottsdale, Arizona
  - Galderma Study Site, Solana Beach, California
  - Galderma Study Site, Bradenton, Florida
  - Galderma Study Site, Austin, Texas
  - Galderma Study Site, Spring, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Investigational Study Product | Reference Product
Started | 59 | 21
Completed | 58 | 21
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational Study Product | Reference Product | Total
Number analyzed (Participants) | 59 | 21 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (10.49) | 51.4 (9.93) | 51.5 (10.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 20 | 76
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 6 | 18
  Not Hispanic or Latino | 47 | 15 | 62
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 59 | 21 | 80
Fitzpatrick Skin Type (FST) [Count of Participants; unit: Participants] — Measure Description: I (White, very fair, red or blond hair, blue eyes, freckles) II (White, fair, red or blond hair; blue, hazel or green eyes) III (Cream white, fair with any eye or hair color, very common) IV (Brown, typical Mediterranean Caucasian skin) V (Dark brown, Middle Eastern skin type) VI (Black)
  Participants
    FST I | 2 | 0 | 2
    FST II | 11 | 6 | 17
    FST III | 25 | 12 | 37
    FST IV | 9 | 2 | 11
    FST V | 9 | 1 | 10
    FST VI | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Wrinkle Assessment Scale (WAS) Score
Description: The WAS is a validated photograph-based outcome instrument that is designed specifically for quantifying facial folds. Scoring of NLF wrinkle severity (grades 0-5, with 0 representing no wrinkles and 5 representing very deep wrinkles, redundant fold) was based on visual live assessment by the Blinded Evaluator at defined timepoints and not on a comparison to the baseline appearance.
  Effectiveness is defined as change from baseline on both sides of the face using WAS at 48 Weeks after the first treatment session.
Time Frame: 48 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Investigational Study Product | Reference Product
Number analyzed (Participants) | 59 | 21
units on a scale
  Left NLF | -1.3 [-1.6 to -1.1] | -1.3 [-1.8 to -0.8]
  Right NLF | -1.2 [-1.4 to -1.0] | -1.3 [-1.8 to -0.9]

2. Secondary Outcome: Change in Wrinkle Assessment Scale (WAS) Score
Description: The WAS is a validated photograph-based outcome instrument that is designed specifically for quantifying facial folds. Scoring of NLF wrinkle severity (grades 0-5, with 0 representing no wrinkles and 5 representing very deep wrinkles, redundant fold) was based on visual live assessment by the Blinded Evaluator at defined timepoints and not on a comparison to the baseline appearance.
  Effectiveness is defined as change from baseline on both sides of the face as assessed by the Blinded Evaluator using WAS at X weeks
Time Frame: Weeks 16, 24, 32, and 40
Population: Intent-to-Treat Population, Observed cases
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Investigational Study Product | Reference Product
Number analyzed (Participants) | 59 | 21
units on a scale
  Week 16- Left NLF: number analyzed (Participants) | 57 | 21
  Week 16- Left NLF | -1.3 (0.96) | -1.5 (0.81)
  Week 16- Right NLF: number analyzed (Participants) | 57 | 21
  Week 16- Right NLF | -1.1 (0.69) | -1.5 (0.60)
  Week 24- Left NLF: number analyzed (Participants) | 58 | 21
  Week 24- Left NLF | -1.2 (0.94) | -1.4 (1.21)
  Week 24- Right NFL: number analyzed (Participants) | 58 | 21
  Week 24- Right NFL | -1.1 (0.84) | -1.5 (0.68)
  Week 32- Left NLF: number analyzed (Participants) | 55 | 21
  Week 32- Left NLF | -1.2 (1.00) | -1.2 (0.93)
  Week 32- Right NLF: number analyzed (Participants) | 55 | 21
  Week 32- Right NLF | -1.1 (0.86) | -1.3 (0.97)
  Week 40- Left NLF | -1.3 (0.94) | -1.4 (0.86)
  Week 40- Right NLF | -1.2 (0.78) | -1.4 (0.80)

3. Secondary Outcome: Responder Rate Based on Global Aesthetic Improvement Scale, Subject Assessment
Description: Responders defined as at least "improved" (improved, much improved, very much improved) as assessed by the subject
Time Frame: Weeks 16, 24, 32, 40, and 48.
Population: Intent-to-Treat Population, observed cases
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Study Product | Reference Product
Number analyzed (Participants) | 59 | 21
Participants
  Week 16: number analyzed (Participants) | 57 | 21
  Week 16 | 54 | 20
  Week 24: number analyzed (Participants) | 58 | 21
  Week 24 | 53 | 20
  Week 32: number analyzed (Participants) | 57 | 21
  Week 32 | 52 | 20
  Week 40 | 51 | 20
  Week 48: number analyzed (Participants) | 58 | 21
  Week 48 | 51 | 21

4. Secondary Outcome: Responder Rate Based on the Global Aesthetic Improvement Scale, Treating Investigator Assessment
Description: Responders defined as at least "improved" (improved, much improved, very much improved) as assessed by the Treating Investigator
Time Frame: Weeks 16, 24, 32, 40 and 48
Population: Intent-to-Treat Population, Observed cases
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Study Product | Reference Product
Number analyzed (Participants) | 59 | 21
Participants
  Week 16: number analyzed (Participants) | 56 | 21
  Week 16 | 56 | 21
  Week 24: number analyzed (Participants) | 58 | 21
  Week 24 | 58 | 21
  Week 32: number analyzed (Participants) | 57 | 21
  Week 32 | 57 | 21
  Week 40 | 59 | 21
  Week 48: number analyzed (Participants) | 57 | 21
  Week 48 | 57 | 21

5. Secondary Outcome: FACE-Q Appraisal of Lines Rasch Transformed Total Scores: NLF Questionnaire
Description: Subjects' satisfaction using the validated FACE-Q Scale, Rasch-transformed total score (0-100) according to the FACE-Q manual; the higher total score indicated greater subject satisfaction
Time Frame: Baseline and at weeks 24, 32, 40 and 48
Population: Intent-to-Treat Population, Observed cases
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Investigational Study Product | Reference Product
Number analyzed (Participants) | 59 | 21
score on a scale
  Baseline | 37.8 (20.89) | 39.4 (16.22)
  Week 24: number analyzed (Participants) | 58 | 21
  Week 24 | 75.3 (23.10) | 81.2 (19.83)
  Week 32 | 72.4 (24.44) | 73.2 (23.80)
  Week 40 | 71.3 (25.31) | 77.2 (21.33)
  Week 48 | 74.3 (23.60) | 79.9 (19.39)

6. Secondary Outcome: Satisfaction With Treatment: Does the Treatment Make You Look Younger?
Description: A 5-point subject satisfaction questionnaire with the following responses: Very Satisfied, Satisfied, Neutral, Dissatisfied, Very Dissatisfied.
Time Frame: Week 16, 24, 32, 40 and 48
Population: ITT- observed cases
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Study Product | Reference Product
Number analyzed (Participants) | 59 | 21
Participants
  Week 16: number analyzed (Participants) | 57 | 21
  Week 16: Very Satisfied | 29 | 11
  Week 16: Satisfied | 19 | 10
  Week 16: Neutral (not satisfied or dissatisfied) | 6 | 0
  Week 16: Dissatisfied | 2 | 0
  Week 16: Very Dissatisfied | 1 | 0
  Week 24: number analyzed (Participants) | 58 | 20
  Week 24: Very Satisfied | 22 | 8
  Week 24: Satisfied | 28 | 12
  Week 24: Neutral (not satisfied or dissatisfied) | 6 | 0
  Week 24: Dissatisfied | 2 | 0
  Week 24: Very Dissatisfied | 0 | 0
  Week 32: number analyzed (Participants) | 57 | 21
  Week 32: Very Satisfied | 25 | 10
  Week 32: Satisfied | 18 | 9
  Week 32: Neutral (not satisfied or dissatisfied) | 12 | 2
  Week 32: Dissatisfied | 2 | 0
  Week 32: Very Dissatisfied | 0 | 0
  Week 40: Very Satisfied | 24 | 11
  Week 40: Satisfied | 26 | 7
  Week 40: Neutral (not satisfied or dissatisfied) | 6 | 3
  Week 40: Dissatisfied | 2 | 0
  Week 40: Very Dissatisfied | 1 | 0
  Week 48: number analyzed (Participants) | 58 | 21
  Week 48: Very Satisfied | 23 | 10
  Week 48: Satisfied | 25 | 9
  Week 48: Neutral (not satisfied or dissatisfied) | 7 | 2
  Week 48: Dissatisfied | 3 | 0
  Week 48: Very Dissatisfied | 0 | 0

7. Secondary Outcome: Subject Satisfaction With Treatment: Does the Treatment Improve Your Attractiveness?
Description: as for outcome 6
Time Frame: Week 16, 24, 32, 40 and 48
Population: ITT- observed cases
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Study Product | Reference Product
Number analyzed (Participants) | 59 | 21
Participants
  Week 16: number analyzed (Participants) | 57 | 21
  Week 16: Very satisfied | 21 | 8
  Week 16: Satisfied | 23 | 12
  Week 16: Neutral (not satisfied or dissatisfied) | 10 | 1
  Week 16: Dissatisfied | 2 | 0
  Week 16: Very Dissatisfied | 1 | 0
  Week 24: number analyzed (Participants) | 58 | 20
  Week 24: Very satisfied | 19 | 8
  Week 24: Satisfied | 25 | 10
  Week 24: Neutral (not satisfied or dissatisfied) | 12 | 2
  Week 24: Dissatisfied | 2 | 0
  Week 24: Very Dissatisfied | 0 | 0
  Week 32: number analyzed (Participants) | 57 | 21
  Week 32: Very satisfied | 25 | 9
  Week 32: Satisfied | 17 | 9
  Week 32: Neutral (not satisfied or dissatisfied) | 13 | 3
  Week 32: Dissatisfied | 2 | 0
  Week 32: Very Dissatisfied | 0 | 0
  Week 40: Very satisfied | 24 | 11
  Week 40: Satisfied | 23 | 6
  Week 40: Neutral (not satisfied or dissatisfied) | 9 | 4
  Week 40: Dissatisfied | 2 | 0
  Week 40: Very Dissatisfied | 1 | 0
  Week 48: number analyzed (Participants) | 58 | 21
  Week 48: Very satisfied | 20 | 9
  Week 48: Satisfied | 24 | 9
  Week 48: Neutral (not satisfied or dissatisfied) | 11 | 3
  Week 48: Dissatisfied | 3 | 0
  Week 48: Very Dissatisfied | 0 | 0

8. Secondary Outcome: Subject Satisfaction With Treatment; Does the Treatment Make You Feel Better About Yourself?
Description: as for outcome 6
Time Frame: Week 16, 24, 32, 40 and 48
Population: ITT- observed cases
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Study Product | Reference Product
Number analyzed (Participants) | 59 | 21
Participants
  Week 16: number analyzed (Participants) | 57 | 21
  Week 16: Very Satisfied | 24 | 11
  Week 16: Satisfied | 19 | 10
  Week 16: Neutral (not satisfied or dissatisfied) | 11 | 0
  Week 16: Dissatisfied | 2 | 0
  Week 16: Very Dissatisfied | 1 | 0
  Week 24: number analyzed (Participants) | 58 | 20
  Week 24: Very Satisfied | 21 | 10
  Week 24: Satisfied | 28 | 10
  Week 24: Neutral (not satisfied or dissatisfied) | 6 | 0
  Week 24: Dissatisfied | 3 | 0
  Week 24: Very Dissatisfied | 0 | 0
  Week 32: number analyzed (Participants) | 57 | 21
  Week 32: Very Satisfied | 27 | 10
  Week 32: Satisfied | 17 | 8
  Week 32: Neutral (not satisfied or dissatisfied) | 12 | 3
  Week 32: Dissatisfied | 1 | 0
  Week 32: Very Dissatisfied | 0 | 0
  Week 40: Very Satisfied | 24 | 13
  Week 40: Satisfied | 21 | 4
  Week 40: Neutral (not satisfied or dissatisfied) | 11 | 4
  Week 40: Dissatisfied | 2 | 0
  Week 40: Very Dissatisfied | 1 | 0
  Week 48: number analyzed (Participants) | 58 | 21
  Week 48: Very Satisfied | 24 | 11
  Week 48: Satisfied | 23 | 7
  Week 48: Neutral (not satisfied or dissatisfied) | 9 | 3
  Week 48: Dissatisfied | 2 | 0
  Week 48: Very Dissatisfied | 0 | 0

9. Secondary Outcome: Subject Satisfaction With Treatment: Does the Treatment Improve Your Self-confidence?
Description: as for outcome 6
Time Frame: Week 16, 24, 32, 40 and 48
Population: ITT- observed cases
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Study Product | Reference Product
Number analyzed (Participants) | 59 | 21
Participants
  Week 16: number analyzed (Participants) | 57 | 21
  Week 16: Very Satisfied | 21 | 7
  Week 16: Satisfied | 19 | 12
  Week 16: Neutral (not satisfied or dissatisfied) | 15 | 2
  Week 16: Dissatisfied | 1 | 0
  Week 16: Very Dissatisfied | 1 | 0
  Week 24: number analyzed (Participants) | 58 | 20
  Week 24: Very Satisfied | 18 | 7
  Week 24: Satisfied | 24 | 8
  Week 24: Neutral (not satisfied or dissatisfied) | 13 | 5
  Week 24: Dissatisfied | 3 | 0
  Week 24: Very Dissatisfied | 0 | 0
  Week 32: number analyzed (Participants) | 57 | 21
  Week 32: Very Satisfied | 24 | 9
  Week 32: Satisfied | 17 | 7
  Week 32: Neutral (not satisfied or dissatisfied) | 14 | 5
  Week 32: Dissatisfied | 2 | 0
  Week 32: Very Dissatisfied | 0 | 0
  Week 40: Very Satisfied | 22 | 11
  Week 40: Satisfied | 20 | 5
  Week 40: Neutral (not satisfied or dissatisfied) | 14 | 5
  Week 40: Dissatisfied | 2 | 0
  Week 40: Very Dissatisfied | 1 | 0
  Week 48: number analyzed (Participants) | 58 | 21
  Week 48: Very Satisfied | 22 | 9
  Week 48: Satisfied | 19 | 8
  Week 48: Neutral (not satisfied or dissatisfied) | 15 | 4
  Week 48: Dissatisfied | 2 | 0
  Week 48: Very Dissatisfied | 0 | 0

10. Secondary Outcome: Subject Satisfaction With Treatment: Does the Treatment Improve Overall Satisfaction With Your Appearance?
Description: as for outcome 6
Time Frame: Week 16, 24, 32, 40 and 48
Population: ITT- observed cases
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Study Product | Reference Product
Number analyzed (Participants) | 59 | 21
Participants
  Week 16: number analyzed (Participants) | 57 | 21
  Week 16: Very Satisfied | 23 | 8
  Week 16: Satisfied | 26 | 12
  Week 16: Neutral | 6 | 1
  Week 16: Dissatisfied | 1 | 0
  Week 16: Very Dissatisfied | 1 | 0
  Week 24: number analyzed (Participants) | 58 | 20
  Week 24: Very Satisfied | 17 | 7
  Week 24: Satisfied | 34 | 13
  Week 24: Neutral | 5 | 0
  Week 24: Dissatisfied | 2 | 0
  Week 24: Very Dissatisfied | 0 | 0
  Week 32: number analyzed (Participants) | 57 | 21
  Week 32: Very Satisfied | 24 | 12
  Week 32: Satisfied | 22 | 8
  Week 32: Neutral | 10 | 1
  Week 32: Dissatisfied | 1 | 0
  Week 32: Very Dissatisfied | 0 | 0
  Week 40: Very Satisfied | 23 | 12
  Week 40: Satisfied | 26 | 6
  Week 40: Neutral | 7 | 3
  Week 40: Dissatisfied | 2 | 0
  Week 40: Very Dissatisfied | 1 | 0
  Week 48: number analyzed (Participants) | 58 | 21
  Week 48: Very Satisfied | 25 | 11
  Week 48: Satisfied | 20 | 8
  Week 48: Neutral | 11 | 2
  Week 48: Dissatisfied | 2 | 0
  Week 48: Very Dissatisfied | 0 | 0

11. Secondary Outcome: Subject Satisfaction With Treatment: Does the Treatment Make You Look/Feel More Confident in Your Life?
Description: as for outcome 6
Time Frame: Week 16, 24, 32, 40 and 48
Population: ITT- observed cases
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Study Product | Reference Product
Number analyzed (Participants) | 59 | 21
Participants
  Week 16: number analyzed (Participants) | 57 | 21
  Week 16: Very Satisfied | 16 | 5
  Week 16: Satisfied | 23 | 11
  Week 16: Neutral (not satisfied or dissatisfied) | 15 | 5
  Week 16: Dissatisfied | 2 | 0
  Week 16: Very Dissatisfied | 1 | 0
  Week 24: number analyzed (Participants) | 58 | 20
  Week 24: Very Satisfied | 16 | 6
  Week 24: Satisfied | 25 | 8
  Week 24: Neutral (not satisfied or dissatisfied) | 15 | 6
  Week 24: Dissatisfied | 2 | 0
  Week 24: Very Dissatisfied | 0 | 0
  Week 32: number analyzed (Participants) | 57 | 21
  Week 32: Very Satisfied | 21 | 8
  Week 32: Satisfied | 16 | 9
  Week 32: Neutral (not satisfied or dissatisfied) | 18 | 4
  Week 32: Dissatisfied | 2 | 0
  Week 32: Very Dissatisfied | 0 | 0
  Week 40: Very Satisfied | 21 | 9
  Week 40: Satisfied | 21 | 7
  Week 40: Neutral (not satisfied or dissatisfied) | 14 | 5
  Week 40: Dissatisfied | 2 | 0
  Week 40: Very Dissatisfied | 1 | 0
  Week 48: number analyzed (Participants) | 58 | 21
  Week 48: Very Satisfied | 21 | 9
  Week 48: Satisfied | 20 | 6
  Week 48: Neutral (not satisfied or dissatisfied) | 15 | 6
  Week 48: Dissatisfied | 2 | 0
  Week 48: Very Dissatisfied | 0 | 0

12. Secondary Outcome: Subject Satisfaction With Treatment: Does the Treatment Make You Look the Way You Feel?
Description: as for outcome 6
Time Frame: Week 16, 24, 32, 40 and 48
Population: ITT- observed cases
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Study Product | Reference Product
Number analyzed (Participants) | 59 | 21
Participants
  Week 16: number analyzed (Participants) | 57 | 21
  Week 16: Very Satisfied | 16 | 5
  Week 16: Satisfied | 25 | 13
  Week 16: Neutral (not satisfied or dissatisfied) | 14 | 3
  Week 16: Dissatisfied | 1 | 0
  Week 16: Very Dissatisfied | 1 | 0
  Week 24: number analyzed (Participants) | 58 | 20
  Week 24: Very Satisfied | 16 | 7
  Week 24: Satisfied | 30 | 10
  Week 24: Neutral (not satisfied or dissatisfied) | 10 | 3
  Week 24: Dissatisfied | 2 | 0
  Week 24: Very Dissatisfied | 0 | 0
  Week 32: number analyzed (Participants) | 57 | 21
  Week 32: Very Satisfied | 21 | 10
  Week 32: Satisfied | 19 | 8
  Week 32: Neutral (not satisfied or dissatisfied) | 14 | 3
  Week 32: Dissatisfied | 3 | 0
  Week 32: Very Dissatisfied | 0 | 0
  Week 40: Very Satisfied | 22 | 11
  Week 40: Satisfied | 21 | 6
  Week 40: Neutral (not satisfied or dissatisfied) | 12 | 4
  Week 40: Dissatisfied | 3 | 0
  Week 40: Very Dissatisfied | 1 | 0
  Week 48: number analyzed (Participants) | 58 | 21
  Week 48: Very Satisfied | 19 | 10
  Week 48: Satisfied | 21 | 4
  Week 48: Neutral (not satisfied or dissatisfied) | 16 | 7
  Week 48: Dissatisfied | 2 | 0
  Week 48: Very Dissatisfied | 0 | 0

13. Secondary Outcome: Subject Satisfaction With Treatment: Does the Treatment Improve Your Facial Symmetry/Balance?
Description: as for outcome 6
Time Frame: Week 16, 24, 32, 40 and 48
Population: ITT- observed cases
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Study Product | Reference Product
Number analyzed (Participants) | 59 | 21
Participants
  Week 16: number analyzed (Participants) | 57 | 21
  Week 16: Very Satisfied | 24 | 9
  Week 16: Satisfied | 21 | 10
  Week 16: Neutral (not satisfied or dissatisfied) | 9 | 2
  Week 16: Dissatisfied | 2 | 0
  Week 16: Very Dissatisfied | 1 | 0
  Week 24: number analyzed (Participants) | 58 | 20
  Week 24: Very Satisfied | 17 | 7
  Week 24: Satisfied | 27 | 10
  Week 24: Neutral (not satisfied or dissatisfied) | 11 | 2
  Week 24: Dissatisfied | 3 | 1
  Week 24: Very Dissatisfied | 0 | 0
  Week 32: number analyzed (Participants) | 57 | 21
  Week 32: Very Satisfied | 22 | 11
  Week 32: Satisfied | 20 | 8
  Week 32: Neutral (not satisfied or dissatisfied) | 11 | 2
  Week 32: Dissatisfied | 4 | 0
  Week 32: Very Dissatisfied | 0 | 0
  Week 40: Very Satisfied | 22 | 10
  Week 40: Satisfied | 26 | 8
  Week 40: Neutral (not satisfied or dissatisfied) | 7 | 3
  Week 40: Dissatisfied | 3 | 0
  Week 40: Very Dissatisfied | 1 | 0
  Week 48: number analyzed (Participants) | 58 | 21
  Week 48: Very Satisfied | 20 | 9
  Week 48: Satisfied | 24 | 9
  Week 48: Neutral (not satisfied or dissatisfied) | 11 | 3
  Week 48: Dissatisfied | 3 | 0
  Week 48: Very Dissatisfied | 0 | 0

14. Secondary Outcome: Subject Satisfaction With Treatment: Would You Say the Subtle Treatment Results Over Time Was Worth it?
Description: A 5-point subject satisfaction questionnaire with the following responses: Strongly Agree, Agree, Neither Agree Nor Disagree, Disagree, Strongly Disagree.
Time Frame: Week 16, 24, 32, 40 and 48
Population: ITT- observed cases
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Study Product | Reference Product
Number analyzed (Participants) | 59 | 21
Participants
  Week 16: number analyzed (Participants) | 57 | 21
  Week 16: Strongly Agree | 37 | 17
  Week 16: Agree | 14 | 4
  Week 16: Neither agree or disagree | 2 | 0
  Week 16: Disagree | 2 | 0
  Week 16: Strongly Disagree | 2 | 0
  Week 24: number analyzed (Participants) | 58 | 20
  Week 24: Strongly Agree | 34 | 14
  Week 24: Agree | 16 | 6
  Week 24: Neither agree or disagree | 4 | 0
  Week 24: Disagree | 3 | 0
  Week 24: Strongly Disagree | 1 | 0
  Week 32: number analyzed (Participants) | 57 | 21
  Week 32: Strongly Agree | 31 | 15
  Week 32: Agree | 15 | 6
  Week 32: Neither agree or disagree | 7 | 0
  Week 32: Disagree | 2 | 0
  Week 32: Strongly Disagree | 2 | 0
  Week 40: Strongly Agree | 31 | 13
  Week 40: Agree | 16 | 5
  Week 40: Neither agree or disagree | 8 | 2
  Week 40: Disagree | 1 | 1
  Week 40: Strongly Disagree | 3 | 0
  Week 48: number analyzed (Participants) | 58 | 21
  Week 48: Strongly Agree | 31 | 15
  Week 48: Agree | 15 | 4
  Week 48: Neither agree or disagree | 8 | 2
  Week 48: Disagree | 3 | 0
  Week 48: Strongly Disagree | 1 | 0

15. Secondary Outcome: Subject Satisfaction With Treatment: Would You Say the Treatment Results Are Natural Looking?
Description: as for outcome 14
Time Frame: Week 16, 24, 32, 40 and 48
Population: ITT- observed cases
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Study Product | Reference Product
Number analyzed (Participants) | 59 | 21
Participants
  Week 16: number analyzed (Participants) | 57 | 21
  Week 16: Strongly Agree | 38 | 17
  Week 16: Agree | 16 | 4
  Week 16: Neither agree or disagree | 2 | 0
  Week 16: Disagree | 1 | 0
  Week 16: Strong Disagree | 0 | 0
  Week 24: number analyzed (Participants) | 58 | 20
  Week 24: Strongly Agree | 38 | 15
  Week 24: Agree | 17 | 5
  Week 24: Neither agree or disagree | 2 | 0
  Week 24: Disagree | 0 | 0
  Week 24: Strong Disagree | 1 | 0
  Week 32: number analyzed (Participants) | 57 | 21
  Week 32: Strongly Agree | 38 | 15
  Week 32: Agree | 16 | 6
  Week 32: Neither agree or disagree | 1 | 0
  Week 32: Disagree | 1 | 0
  Week 32: Strong Disagree | 1 | 0
  Week 40: Strongly Agree | 39 | 14
  Week 40: Agree | 15 | 7
  Week 40: Neither agree or disagree | 4 | 0
  Week 40: Disagree | 0 | 0
  Week 40: Strong Disagree | 1 | 0
  Week 48: number analyzed (Participants) | 58 | 21
  Week 48: Strongly Agree | 36 | 15
  Week 48: Agree | 18 | 5
  Week 48: Neither agree or disagree | 3 | 1
  Week 48: Disagree | 1 | 0
  Week 48: Strong Disagree | 0 | 0

16. Secondary Outcome: Subject Satisfaction With Treatment: Would You do the Treatment Again?
Description: A subject satisfaction question with responses Yes or No.
Time Frame: Week 16, 24, 32, 40 and 48
Population: ITT- observed cases
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Study Product | Reference Product
Number analyzed (Participants) | 59 | 21
Participants
  Week 16: number analyzed (Participants) | 57 | 21
  Week 16: Yes | 53 | 19
  Week 16: No | 4 | 2
  Week 24: number analyzed (Participants) | 58 | 20
  Week 24: Yes | 54 | 17
  Week 24: No | 4 | 3
  Week 32: number analyzed (Participants) | 57 | 21
  Week 32: Yes | 50 | 18
  Week 32: No | 7 | 3
  Week 40: Yes | 48 | 18
  Week 40: No | 11 | 3
  Week 48: number analyzed (Participants) | 58 | 21
  Week 48: Yes | 52 | 17
  Week 48: No | 6 | 4

17. Secondary Outcome: Subject Satisfaction With Treatment: Would You Recommend the Treatment to a Friend?
Description: A subject satisfaction question with responses Yes or No.
Time Frame: Week 16, 24, 32, 40 and 48
Population: ITT- observed cases
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Study Product | Reference Product
Number analyzed (Participants) | 59 | 21
Participants
  Week 16: number analyzed (Participants) | 57 | 21
  Week 16: Yes | 52 | 21
  Week 16: No | 5 | 0
  Week 24: number analyzed (Participants) | 58 | 20
  Week 24: Yes | 53 | 20
  Week 24: No | 5 | 0
  Week 32: number analyzed (Participants) | 57 | 21
  Week 32: Yes | 48 | 20
  Week 32: No | 9 | 1
  Week 40: Yes | 51 | 19
  Week 40: No | 8 | 2
  Week 48: number analyzed (Participants) | 58 | 21
  Week 48: Yes | 50 | 19
  Week 48: No | 8 | 2

18. Secondary Outcome: Earliest Time the Subject Reported Feeling Comfortable Returning to Social Engagement Based on Subject Diary Reporting
Description: Subjects were asked to complete the following questions in the subject diary:
  * Did you feel comfortable to return to social engagement today? (Yes or No)
  * If yes, what was the earliest time you felt comfortable to return to social engagement? (Record date and time [using 24-hour clock])
Time Frame: time in hours from treatment procedure after treatments 1,2,3 and 4 at weeks 0, 4, 8, and 12
Population: Intent-to-Treat Population
Measure: Median (Inter-Quartile Range); unit: time in hours
Arm/Group | Investigational Study Product | Reference Product
Number analyzed (Participants) | 59 | 21
time in hours
  After treatment 1 | 1.4 [0.6 to 3.8] | 2 [0.8 to 3.8]
  After treatment 2: number analyzed (Participants) | 58 | 21
  After treatment 2 | 1.6 [0.9 to 4.6] | 1 [0.7 to 3.1]
  After treatment 3: number analyzed (Participants) | 54 | 20
  After treatment 3 | 1.5 [0.8 to 4.2] | 1.5 [0.9 to 7.9]
  After treatment 4: number analyzed (Participants) | 41 | 15
  After treatment 4 | 1.5 [0.9 to 3.4] | 1.0 [0.8 to 3.5]

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Investigational Study Product | Reference Product
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/21
Serious Adverse Events (participants affected / at risk) | 2/59 | 0/21
Other Adverse Events (participants affected / at risk) | 7/59 | 7/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Study Product (N=59) | Reference Product (N=21)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) — right eye
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Study Product (N=59) | Reference Product (N=21)
Hypoesthesia oral (Gastrointestinal disorders) | 1 (1) | 1 (1) — related
Oral disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) — related
Injection site hypoaesthesia (General disorders) | 1 (6) | 0 (0) — related
Injection site paraesthesia (General disorders) | 1 (4) | 0 (0) — related
Injection site induration (General disorders) | 1 (1) | 0 (0) — related
Injection site nodule (General disorders) | 0 (0) | 1 (1) — related
Injection site pain (General disorders) | 0 (0) | 1 (1) — related
Swelling (General disorders) | 0 (0) | 1 (1) — related
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) — related
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) — related
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — related
Headache (Nervous system disorders) | 1 (1) | 2 (3) — related
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — related
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — related
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — related
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — related
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs agree not to present or publish any data or reports collected individually or by subgroup of sites prior to full, initial publication based on all data obtained from all sites

DOCUMENTS (2):
  • Study Protocol (2019-02-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT03780244/Prot_002.pdf
  • Statistical Analysis Plan (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT03780244/SAP_003.pdf